CLINICAL TRIAL: NCT04091009
Title: Effect of Standard of Care Reduced Dose Versus Full Dose Buprenorphine/Naloxone in the Perioperative Period on Pain and Opioid Use Disorder Symptoms
Brief Title: Effect of Standard of Care Reduced Dose Versus Full Dose Buprenorphine/Naloxone in the Perioperative Period on Pain Control and Post-Operative Opioid Use Disorder Symptoms
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi Zhang, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P001092
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Opioid-use Disorder; Opioid Use Disorder, Mild
MeSH Terms: conditions — Opioid-Related Disorders; Lymphoma, Follicular | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continue Group (Active Comparator): Those who continue taking their standard dose of buprenorphine before, during and after surgery.
  Interventions: Drug: Buprenorphine/naloxone
- Reduce Group (Active Comparator): Those who are placed on a lower dose of buprenorphine starting one day before surgery and during the time period after surgery until the pain from the surgery has decreased. Once the pain from the surgery has decreased, you will be put back on your full dose of buprenorphine.
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Participants will be prescribed 8mg buprenorphine daily from the day of surgery until transitioned back to their regular dose of buprenorphine when postoperative surgical pain has subsided

SUMMARY:
The purpose of this research study is to compare two ways of managing pain in people who are taking buprenorphine and are scheduled to undergo surgery. Buprenorphine (subutex) and buprenorphine/naloxone (suboxone) are effective long-term treatments for substance use disorders. The management of pain after surgery in adults taking buprenorphine can be challenging, as buprenorphine may interfere with the effectiveness of other medications used to treat pain.

The investigators want to compare how well pain is managed after surgery ("post-op") in two groups:

The "Continue Group": those who continue taking their standard dose of buprenorphine before, during and after surgery.

The "Reduce Group": those who are placed on a lower dose of buprenorphine starting one day before surgery and during the time period after surgery until the pain from the surgery has decreased. Once the pain from the surgery has decreased, participants will be put back on their full dose of buprenorphine.

The investigators also want to find out if there is a difference in pain, opioid cravings, and relapse rates in the month following surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) health class I-III
* Currently taking buprenorphine or buprenorphine/naloxone daily at a dose of at least 16mg per day for at least the prior 30 days for treatment of Opioid Use Disorder by Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria
* Scheduled for surgery at Massachusetts General Hospital where greater than 3/10 pain is expected on post-operative day 1

Exclusion Criteria:

* Participants unable to consent to the study
* Renal insufficency with a glomerular filtration rate <30ml/min (participants would be unable to use ketorolac which is a part of the multimodal anesthetic plan)
* Liver cirrhosis with a Model for End-Stage Liver Disease (MELD) score > 25 (participants would be unable to use Tylenol which is part of the multimodal anesthetic plan)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain scores at 24 hours post-operative procedure | 24 hours
  Average pain scores at 24 hours post-op

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yi, MD PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No